CLINICAL TRIAL: NCT04505774
Title: A Multicenter, Adaptive, Randomized Controlled Platform Trial of the Safety and Efficacy of Antithrombotic and Additional Strategies in Hospitalized Adults With COVID-19
Brief Title: Accelerating COVID-19 Therapeutic Interventions and Vaccines 4 ACUTE
Acronym: ACTIV-4A
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Matthew Neal MD (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor-Investigator, Matthew Neal MD, MD, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ACTIV-4 ACUTE; 1OT2HL156812-01 (NIH); NCT04359277 (obsolete NCT alias)
Record Dates: First submitted 2020-08-06; First posted 2020-08-10 (Actual); Results first posted 2024-12-30 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Covid19
Keywords: anti-coagulation; antithrombosis; anticoagulation; ACTIV; inpatient; heparin; p2y12; endothelial dysfunction; vascular integrity; P-selectin; crizanlizumab; SGLT-2 inhibitor
MeSH Terms: conditions — COVID-19 | interventions — Heparin; Enoxaparin; Dalteparin; Tinzaparin; Ticagrelor; Prasugrel Hydrochloride; Clopidogrel; crizanlizumab; Sodium-Glucose Transporter 2 Inhibitors; dapagliflozin; empagliflozin; Canagliflozin; ertugliflozin

STUDY DESIGN:
Intervention Model Description: This is an adaptive design
Masking Description: There will be independent masked adjudicators.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (8):
- Therapeutic Dose Anticoagulation (Other): increased dose of heparin above standard of care.
  1.0 - This arm was stopped in severe patients in December 2020 and results are published in PMID: 34351722 (NEJM, August, 2021) (see reference section for citation). This arm was stopped for moderate patients in January 2021.
  Interventions: Drug: theraputic heparin
- Prophylactic Dose Anticoagulation (Other): Heparin standard of care
  1.0 - this arm was stopped for all patients in January, 2021 and results are published in PMID: 34351721 (NEJM, August, 2021) (see reference section for citation)
  Interventions: Drug: prophylactic heparin
- Therapeutic Dose Anticoagulation + P2Y12 inhibitor (Other): increased dose of heparin above standard of care with an added P2Y12 inhibitor
  This Arm enrolled moderate illness patients only. Enrollment of moderate illness patients in the trial was ended per DSMB on June 19, 2021 and results are published in PMID: PMID: 35040887 (JAMA, January, 2022) (see reference section for citation)
  Interventions: Drug: theraputic heparin; Drug: P2Y12
- Prophylactic Dose Anticoagulation + P2Y12 inhibitor (Other): Heparin standard of care with an added P2Y12 inhibitor
  This Arm enrolled severe illness patients only. Enrollment of severe illness patients in the trial was ended per DSMB in June 2022.
  Interventions: Drug: prophylactic heparin; Drug: P2Y12
- Standard of Care + Crizanlizumab (Other): Standard of care plus crizanlizumab infusion
  This arm will enroll moderate and severe illness patients
  This arm was ended for all patients per the DSMB in September 2022.
  Interventions: Drug: Crizanlizumab Injection
- Standard of Care + SGLT2 inhibitor (Other): Standard of care plus SGLT2 inhibitor
  This arm will enroll moderate and severe illness patients
  This arm was ended in March 2023
  Interventions: Drug: SGLT2 inhibitor
- Standard of Care (SGLT2 arm) (Other): Standard of care only
  This arm will enroll moderate and severe illness patients
  This arm was ended in March 2023
  Interventions: Drug: SGLT2 inhibitor
- Standard of Care (Criza) (Other): Standard of care only This arm will enroll moderate and severe illness patients
  This arm was ended for all patients per the DSMB in September 2022.
  Interventions: Drug: Crizanlizumab Injection

INTERVENTIONS:
Drug: theraputic heparin — increased dose of heparin above standard of care.
  Other Names: unfractionated heparin; Enoxaparin; Dalteparin; Tinzaparin; Heparin
  Arms: Therapeutic Dose Anticoagulation; Therapeutic Dose Anticoagulation + P2Y12 inhibitor
Drug: prophylactic heparin — standard of care dose of heparin
  Other Names: enoxaparin; dalteparin; Tinzaparin; Fondparinux; Heparin
  Arms: Prophylactic Dose Anticoagulation; Prophylactic Dose Anticoagulation + P2Y12 inhibitor
Drug: P2Y12 — added P2Y12 inhibitor
  Other Names: Ticagrelor; Prasugrel; Clopidogrel
  Arms: Prophylactic Dose Anticoagulation + P2Y12 inhibitor; Therapeutic Dose Anticoagulation + P2Y12 inhibitor
Drug: Crizanlizumab Injection — crizanlizumab injection
  Arms: Standard of Care (Criza); Standard of Care + Crizanlizumab
Drug: SGLT2 inhibitor — sglt2 inhibitor
  Other Names: dapagliflozin; empagliflozin; canagliflozin; ertugliflozin
  Arms: Standard of Care (SGLT2 arm); Standard of Care + SGLT2 inhibitor

SUMMARY:
This is a randomized, open label, adaptive platform trial to compare the effectiveness of antithrombotic and additional strategies for prevention of adverse outcomes in COVID-19 positive inpatients

DETAILED DESCRIPTION:
The severe acute respiratory syndrome coronavirus 2, which causes the highly contagious coronavirus disease 2019 (COVID-19), has resulted in a global pandemic.

The clinical spectrum of COVID-19 infection is broad, encompassing asymptomatic infection, mild upper respiratory tract illness, and severe viral pneumonia with respiratory failure and death. The risk of thrombotic complications is increased, even as compared to other viral respiratory illnesses, such as influenza. A pro-inflammatory cytokine response as well as induction of procoagulant factors associated with COVID-19 has been proposed to contribute to thrombosis as well as plaque rupture through local inflammation. Patients with COVID-19 are at increased risk for arterial and vein thromboembolism, with high rates observed despite thromboprophylaxis. Autopsy reports have noted micro and macro vascular thrombosis across multiple organ beds consistent with an early hypercoagulable state.

Notably, in COVID-19, data in the U.K. and U.S. document that infection and outcomes of infection are worse in African and Hispanic descent persons than in other groups. The reasons for this are uncertain.

Viral Infection and Thrombosis A large body of literature links inflammation and coagulation; altered hemostasis is a known complication of respiratory viral infections. Procoagulant markers are severely elevated in viral infections. Specifically, proinflammatory cytokines in viral infections upregulate expression of tissue factor, markers of thrombin generation, platelet activation, and down-regulate natural anticoagulant proteins C and S.

Studies have demonstrated significant risk of deep venous thrombosis (DVT), pulmonary embolism (PE), and myocardial infarction (MI) associated with viral respiratory infections. In a series of patients with fatal influenza H1N1, 75% had pulmonary thrombi on autopsy (a rate considerably higher than reported on autopsy studies among the general intensive care unit population). Incidence ratio for acute myocardial infarction in the context of Influenza A is over 10. Severe acute respiratory syndrome coronavirus-1 (SARS CoV-1) and influenza have been associated with disseminated intravascular coagulation (DIC), endothelial damage, DVT, PE, and large artery ischemic stroke. Patients with Influenza H1N1 and acute respiratory distress syndrome (ARDS) had a 23.3-fold higher risk for pulmonary embolism, and a 17.9-fold increased risk for deep vein thrombosis. Compared to those treated with systemic anticoagulation, those without treatment were 33 times more likely to suffer a VTE.

Thrombosis, both microvascular and macrovascular, is a prominent feature in multiple organs at autopsy in fatal cases of COVID-19. Thrombosis may thus contribute to respiratory failure, renal failure, and hepatic injury in COVID-19. The number of megakaryocytes in tissues is higher than in other forms of ARDS, and thrombi are platelet-rich based on specific staining. Thrombotic stroke has been reported in young COVID-19 patients with no cardiovascular risk factors. Both arterial and venous thrombotic events have been seen in increasing numbers of hospitalized patients infected with COVID-19. The incidence of thrombosis has ranged from 10 to 30% in hospitalized patients; however, this varies by type of thrombosis captured (arterial or vein) and severity of illness (ICU level care, requiring mechanical ventilation, etc.).

Additional treatment strategies Data from the multiplatform randomized controlled trial (mpRCT) demonstrated that (1) therapeutic dose anticoagulation with heparin was not beneficial in improving clinical outcomes compared to standard of care prophylactic dose heparin in severely ill (ICU level of care) patients, and (2) therapeutic dose anticoagulation with heparin was beneficial in improving organ support free days compared to standard of care prophylactic dose heparin in moderately ill (hospitalized and not requiring organ support) patients. However, there remains significant residual risk for adverse clinical outcomes and excess mortality for severely ill as well as moderately ill patients.

Antithrombotic regimens that are shown to be efficacious will be combined in clinical practice with other agents to treat COVID-19 hospitalized patients. This adaptive platform trial will test other promising agents when added to proven therapies, such as heparin. The rationale and risks for each agent will be included in the arm-specific appendix. Two specific agents to be added as arms, effective October 2021, include the P-selectin inhibitor, Crizanlizumab as well as SGLT2 inhibitors. P-selectin may play a proximal role in the inflammatory and thrombotic cascade in patients with COVID-19 and P-selectin inhibition may be a effective in preventing downstream sequelae. In addition, SGLT-2 inhibitors have been shown to decrease capillary leak and may promote vascular integrity in COVID-19.

This platform trial will have multiple arms, which may be dropped or added as the platform trial progresses. Sample size will be flexible: the trial will be stopped for efficacy or futility based on pre-determined statistical thresholds as defined in the arm-specific appendices. Each arm will have an adaptive component for determinations of futility or success.

Randomization assignments are at the participant level, stratified by enrolling site and by ICU level of care vs non-ICU level of care and/or other arm-specific criteria.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Hospitalized for COVID-19
* Enrolled within 72 hours of hospital admittance or 72 hours of positive COVID test
* Expected to require hospitalization for > 72 hours

Exclusion Criteria:

* Imminent death
* Requirement for chronic mechanical ventilation via tracheostomy prior to hospitalization
* Pregnancy

Inclusion Criteria for Arm E

Inclusion criteria contained in the master protocol in addition to the following:

Moderate illness severity - defined as non-ICU level of care at the time of randomization (not receiving high flow nasal oxygen (HFNO), non-invasive ventilation (NIV), invasive ventilation (IV), vasopressors or inotropes, or extracorporeal membrane oxygenation (ECMO) OR Severe illness severity - defined as ICU level of care at the time of randomization (receiving HFNO, NIV, IV, vasopressors or inotropes, or ECMO)

For moderate illness severity, participants are required to meet one or more of the following risk criteria:

1. Age ≥ 65 years or
2. ≥2 of the following -

   * O2 supplementation > 2 liters per minute
   * BMI ≥ 35
   * GFR ≤ 60
   * History of Type 2 diabetes
   * History of heart failure (regardless of ejection fraction)
   * D dimer ≥ 2x the site's upper limit of normal (ULN)
   * Troponin ≥ 2x the site's ULN
   * BNP≥100 pg/mL or NT-proBNP≥300 pg/mL
   * CRP ≥50 mg/L

Exclusion Criteria for Arm E

* Exclusion criteria contained in the master protocol, and
* Any condition that, in the opinion of the investigator, precludes the use of crizanlizumab such as uncontrolled bleeding or severe anemia (hemoglobin<4 g/dL)
* Open label treatment with crizanlizumab within the past three months

Inclusion Criteria for Arm F

Inclusion criteria contained in the master protocol in addition to the following:

Moderate illness severity - defined as non-ICU level of care at the time of randomization (not receiving high flow nasal oxygen (HFNO), non-invasive ventilation (NIV), invasive ventilation (IV), vasopressors or inotropes, or extracorporeal membrane oxygenation (ECMO)) OR Severe illness severity - defined as ICU level of care at the time of randomization (receiving HFNO, NIV, IV, vasopressors or inotropes, or ECMO)

For moderate illness severity, participants are required to meet one or more of the following risk criteria:

1. Age ≥ 65 years or
2. ≥2 of the following-

   * O2 supplementation > 2 liters per minute
   * BMI ≥ 35
   * GFR ≤ 60
   * History of Type 2 diabetes
   * History of heart failure (regardless of ejection fraction)
   * D dimer ≥ 2x the site's upper limit of normal (ULN)
   * Troponin ≥ 2x the site's ULN
   * BNP≥100 pg/mL or NT-proBNP≥300 pg/mL
   * CRP ≥50 mg/L

Exclusion Criteria for Arm F

In addition to the exclusion criteria noted in the master protocol, arm-specific exclusion criteria are as follows:

* Known hypersensitivity to any SGLT2 inhibitors
* Type 1 diabetes
* History of diabetic ketoacidosis
* eGFR <20 and/or requirement for renal replacement therapy
* Open label treatment with any SGLT2 inhibitor

  * Based on a recommendation from the ACTIV4 DSMB on December 19, 2020, enrollment of patients requiring ICU level of care into the therapeutic anti-coagulation arm was stopped due to meeting a futility threshold and a potential for harm for this sub-group could not be excluded. Enrollment continues for moderately ill hospitalized COVID-19 patients.
  * Based on a recommendation from the ACTIV4 DSMB on June 18, 2021, enrollment of patients not requiring ICU level of care and randomized to P2Y12 or standard care was stopped due to meeting a futility threshold. Enrollment continues for severely ill (ICU level of care) hospitalized COVID-19 patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3591 (Actual)
Dates: Start 2020-09-04 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2024-01-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judith Hochman, MD, Study Chair — NYU Langone Health; Scott Solomon, MD, Principal Investigator — Brigham and Women's Hospital; Mikhail Kosiborod, MD, Principal Investigator — Saint Lukes; Jeffrey Berger, MD, Principal Investigator — NYU Langone Health; MATTHEW D NEAL, MD, Study Chair — University of Pittsburgh
Locations (100):
- United States (80):
  - University of Alabama, Birmingham, Alabama
  - University of Arizona, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Kaiser Permanente Fontana, Fontana, California
  - Kaiser Permanente Los Angeles, Los Angeles, California
  - Smidt Heart Institute at Cedars-Sinai, Los Angeles, California
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - UC San Diego Hillcrest, San Diego, California
  - Zuckerberg San Francisco General Hospital, San Francisco, California
  - UCSF San Francisco, San Francisco, California
  - Stanford University Medical Center, Stanford, California
  - Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center, Torrance, California
  - Denver Health and Hospital Authority, Denver, Colorado
  - St. Mary's Hospital & Regional Medical Center, Grand Junction, Colorado
  - Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - University of Florida, Gainesville, Florida
  - Memorial Hospital, Jacksonville, Florida
  - AdventHealth Tampa, Tampa, Florida
  - Emory, Atlanta, Georgia
  - Morehouse School of Medicine, Atlanta, Georgia
  - Queens Medical Center, Honolulu, Hawaii
  - Memorial Hospital, Belleville, Illinois
  - Cook County Health, Chicago, Illinois
  - University of Illinois at Chicago Health (UIH), Chicago, Illinois
  - OSF Little Company of Mary Medical Center (OSF LCM), Evergreen Park, Illinois
  - Indiana University Health Methodist Hospital, Indianapolis, Iowa
  - Kansas University Medical Center, Kansas City, Kansas
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Boston University, Boston, Massachusetts
  - St Elizabeth's Medical Center, Brighton, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - University of Massachusetts, Worcester, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Wayne State University, Detroit, Michigan
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Washington University School of Medicine, ACCS Research, St Louis, Missouri
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Cooper Health, Camden, New Jersey
  - Englewood Health, Englewood, New Jersey
  - Atlantic Health System, Morristown, New Jersey
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - AtlantiCare Regional Medical Center, Pomona, New Jersey
  - Albany Medical College, Albany, New York
  - Mercy Hospital Buffalo, Buffalo, New York
  - VA New York Harbor Healthcare System, New York, New York
  - NYU Langone, New York, New York
  - Mt. Sinai Hospital, New York, New York
  - SUNY Upstate University Hospital, Syracuse, New York
  - Jacobi Medical Center, The Bronx, New York
  - Montefiore Medical Center, The Bronx, New York
  - Westchester Medical Center, Valhalla, New York
  - Duke University Hospital, Durham, North Carolina
  - Wake Forest, Winston-Salem, North Carolina
  - Cleveland Clinic Akron General, Akron, Ohio
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - The MetroHealth System, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State Universtiy Wexner Medical Center, Columbus, Ohio
  - Mercy Health St Vincent Medical Center, Toledo, Ohio
  - Ascension St. John Clinical Research Institute, Tulsa, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - Geisinger Research, Danville, Pennsylvania
  - Doylestown Cardiology Associates, Doylestown, Pennsylvania
  - Penn State Health Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Temple University, Philadelphia, Pennsylvania
  - UPMC Presbyterian, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - The Miriam Hospital, Providence, Rhode Island
  - Sarah Cannon and HCA Research Institute, Nashville, Tennessee
  - Skyline Medical Center, Nashville, Tennessee
  - University of Texas at Austin, Austin, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Medical City Ft Worth, Fort Worth, Texas
  - Baylor Scott and White Medical Center - Temple, Temple, Texas
  - HCA Henrico Doctors Hospital, Richmond, Virginia
  - Swedish Hospital, Seattle, Washington
  - West Virginia University CTR, Morgantown, West Virginia
  - University of Wisconsin Hospital; Meriter Hospital (UW affiliated), Madison, Wisconsin
- Brazil (6):
  - Hospital Universitario Sao Francisco de Assis, Bragança Paulista
  - União Brasileira de Educação e Assistência - Hospital São Lucas da PUCRS, Porto Alegre
  - Centro de Estudos Clínicos do Hospital Cárdio Pulmonar, Salvador
  - Fundação Faculdade Regional De Medicina De São José Do Rio Preto, São José do Rio Preto
  - Instituto Dante Pazzanese de Cardiologia, São Paulo
  - Instituto do Coração do Hospital das Clínicas da Faculdade de Medicina da USP-InCor-HCFMUSP, São Paulo
- Italy (7):
  - Azienda Ospedaliero Sant Anna e San Sebastiano, Caserta
  - Maria Cecilia Hospital , Cotignola, Ravenna, Cotignola
  - Università degli Studi di Ferrara, Ferrara, Ferrara
  - Azienda Ospedaliero -Universitaria Careggi, Florence
  - Policlinico di Napoli, Napoli, Napoli
  - AOU Policlinico di Palermo, Palermo, Palermo
  - ASL-1 Imperiese, Sanremo, Sanremo
- Spain (7):
  - Hospital Universitario A Coruna, A Coruña
  - Hospital Virgen del Mar, Almería
  - Hospital Arnau de Vilanova, Lleida
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Ramon Y Cajal, Madrid
  - Hospital Clínico Universitario de Salamanca, Salamanca
  - Hospital Clínico Universitario de Santiago de Compostela, Santiago de Compostela

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared as per NIH guidelines.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Background] Bikdeli B, Madhavan MV, Jimenez D, Chuich T, Dreyfus I, Driggin E, Nigoghossian C, Ageno W, Madjid M, Guo Y, Tang LV, Hu Y, Giri J, Cushman M, Quere I, Dimakakos EP, Gibson CM, Lippi G, Favaloro EJ, Fareed J, Caprini JA, Tafur AJ, Burton JR, Francese DP, Wang EY, Falanga A, McLintock C, Hunt BJ, Spyropoulos AC, Barnes GD, Eikelboom JW, Weinberg I, Schulman S, Carrier M, Piazza G, Beckman JA, Steg PG, Stone GW, Rosenkranz S, Goldhaber SZ, Parikh SA, Monreal M, Krumholz HM, Konstantinides SV, Weitz JI, Lip GYH; Global COVID-19 Thrombosis Collaborative Group, Endorsed by the ISTH, NATF, ESVM, and the IUA, Supported by the ESC Working Group on Pulmonary Circulation and Right Ventricular Function. COVID-19 and Thrombotic or Thromboembolic Disease: Implications for Prevention, Antithrombotic Therapy, and Follow-Up: JACC State-of-the-Art Review. J Am Coll Cardiol. 2020 Jun 16;75(23):2950-2973. doi: 10.1016/j.jacc.2020.04.031. Epub 2020 Apr 17. PMID 32311448
- [Background] Klok FA, Kruip MJHA, van der Meer NJM, Arbous MS, Gommers DAMPJ, Kant KM, Kaptein FHJ, van Paassen J, Stals MAM, Huisman MV, Endeman H. Incidence of thrombotic complications in critically ill ICU patients with COVID-19. Thromb Res. 2020 Jul;191:145-147. doi: 10.1016/j.thromres.2020.04.013. Epub 2020 Apr 10. PMID 32291094
- [Background] Middeldorp S, Coppens M, van Haaps TF, Foppen M, Vlaar AP, Muller MCA, Bouman CCS, Beenen LFM, Kootte RS, Heijmans J, Smits LP, Bonta PI, van Es N. Incidence of venous thromboembolism in hospitalized patients with COVID-19. J Thromb Haemost. 2020 Aug;18(8):1995-2002. doi: 10.1111/jth.14888. Epub 2020 Jul 27. PMID 32369666
- [Background] Poissy J, Goutay J, Caplan M, Parmentier E, Duburcq T, Lassalle F, Jeanpierre E, Rauch A, Labreuche J, Susen S; Lille ICU Haemostasis COVID-19 Group. Pulmonary Embolism in Patients With COVID-19: Awareness of an Increased Prevalence. Circulation. 2020 Jul 14;142(2):184-186. doi: 10.1161/CIRCULATIONAHA.120.047430. Epub 2020 Apr 24. No abstract available. PMID 32330083
- [Background] Zhou F, Yu T, Du R, Fan G, Liu Y, Liu Z, Xiang J, Wang Y, Song B, Gu X, Guan L, Wei Y, Li H, Wu X, Xu J, Tu S, Zhang Y, Chen H, Cao B. Clinical course and risk factors for mortality of adult inpatients with COVID-19 in Wuhan, China: a retrospective cohort study. Lancet. 2020 Mar 28;395(10229):1054-1062. doi: 10.1016/S0140-6736(20)30566-3. Epub 2020 Mar 11. PMID 32171076
- [Background] Tang N, Bai H, Chen X, Gong J, Li D, Sun Z. Anticoagulant treatment is associated with decreased mortality in severe coronavirus disease 2019 patients with coagulopathy. J Thromb Haemost. 2020 May;18(5):1094-1099. doi: 10.1111/jth.14817. Epub 2020 Apr 27. PMID 32220112
- [Background] Wang L, Zhao L, Li F, Liu J, Zhang L, Li Q, Gu J, Liang S, Zhao Q, Liu J, Xu JF. Risk assessment of venous thromboembolism and bleeding in COVID-19 patients. Clin Respir J. 2022 Mar;16(3):182-189. doi: 10.1111/crj.13467. Epub 2022 Jan 21. PMID 35060325
- [Background] Danzi GB, Loffi M, Galeazzi G, Gherbesi E. Acute pulmonary embolism and COVID-19 pneumonia: a random association? Eur Heart J. 2020 May 14;41(19):1858. doi: 10.1093/eurheartj/ehaa254. No abstract available. PMID 32227120
- [Background] Xie Y, Wang X, Yang P, Zhang S. COVID-19 Complicated by Acute Pulmonary Embolism. Radiol Cardiothorac Imaging. 2020 Mar 16;2(2):e200067. doi: 10.1148/ryct.2020200067. eCollection 2020 Apr. No abstract available. PMID 33778561
- [Background] Beristain-Covarrubias N, Perez-Toledo M, Thomas MR, Henderson IR, Watson SP, Cunningham AF. Understanding Infection-Induced Thrombosis: Lessons Learned From Animal Models. Front Immunol. 2019 Nov 5;10:2569. doi: 10.3389/fimmu.2019.02569. eCollection 2019. PMID 31749809
- [Background] Clayton TC, Gaskin M, Meade TW. Recent respiratory infection and risk of venous thromboembolism: case-control study through a general practice database. Int J Epidemiol. 2011 Jun;40(3):819-27. doi: 10.1093/ije/dyr012. Epub 2011 Feb 15. PMID 21324940
- [Background] Goeijenbier M, van Wissen M, van de Weg C, Jong E, Gerdes VE, Meijers JC, Brandjes DP, van Gorp EC. Review: Viral infections and mechanisms of thrombosis and bleeding. J Med Virol. 2012 Oct;84(10):1680-96. doi: 10.1002/jmv.23354. PMID 22930518
- [Background] Smeeth L, Cook C, Thomas S, Hall AJ, Hubbard R, Vallance P. Risk of deep vein thrombosis and pulmonary embolism after acute infection in a community setting. Lancet. 2006 Apr 1;367(9516):1075-1079. doi: 10.1016/S0140-6736(06)68474-2. PMID 16581406
- [Background] Harms PW, Schmidt LA, Smith LB, Newton DW, Pletneva MA, Walters LL, Tomlins SA, Fisher-Hubbard A, Napolitano LM, Park PK, Blaivas M, Fantone J, Myers JL, Jentzen JM. Autopsy findings in eight patients with fatal H1N1 influenza. Am J Clin Pathol. 2010 Jul;134(1):27-35. doi: 10.1309/AJCP35KOZSAVNQZW. PMID 20551263
- [Background] Kwong JC, Schwartz KL, Campitelli MA, Chung H, Crowcroft NS, Karnauchow T, Katz K, Ko DT, McGeer AJ, McNally D, Richardson DC, Rosella LC, Simor A, Smieja M, Zahariadis G, Gubbay JB. Acute Myocardial Infarction after Laboratory-Confirmed Influenza Infection. N Engl J Med. 2018 Jan 25;378(4):345-353. doi: 10.1056/NEJMoa1702090. PMID 29365305
- [Background] Wong RS, Wu A, To KF, Lee N, Lam CW, Wong CK, Chan PK, Ng MH, Yu LM, Hui DS, Tam JS, Cheng G, Sung JJ. Haematological manifestations in patients with severe acute respiratory syndrome: retrospective analysis. BMJ. 2003 Jun 21;326(7403):1358-62. doi: 10.1136/bmj.326.7403.1358. PMID 12816821
- [Background] Obi AT, Tignanelli CJ, Jacobs BN, Arya S, Park PK, Wakefield TW, Henke PK, Napolitano LM. Empirical systemic anticoagulation is associated with decreased venous thromboembolism in critically ill influenza A H1N1 acute respiratory distress syndrome patients. J Vasc Surg Venous Lymphat Disord. 2019 May;7(3):317-324. doi: 10.1016/j.jvsv.2018.08.010. Epub 2018 Nov 23. PMID 30477976
- [Background] Rapkiewicz AV, Mai X, Carsons SE, Pittaluga S, Kleiner DE, Berger JS, Thomas S, Adler NM, Charytan DM, Gasmi B, Hochman JS, Reynolds HR. Megakaryocytes and platelet-fibrin thrombi characterize multi-organ thrombosis at autopsy in COVID-19: A case series. EClinicalMedicine. 2020 Jun 25;24:100434. doi: 10.1016/j.eclinm.2020.100434. eCollection 2020 Jul. PMID 32766543
- [Background] Oxley TJ, Mocco J, Majidi S, Kellner CP, Shoirah H, Singh IP, De Leacy RA, Shigematsu T, Ladner TR, Yaeger KA, Skliut M, Weinberger J, Dangayach NS, Bederson JB, Tuhrim S, Fifi JT. Large-Vessel Stroke as a Presenting Feature of Covid-19 in the Young. N Engl J Med. 2020 May 14;382(20):e60. doi: 10.1056/NEJMc2009787. Epub 2020 Apr 28. No abstract available. PMID 32343504
- [Background] Al-Samkari H, Karp Leaf RS, Dzik WH, Carlson JCT, Fogerty AE, Waheed A, Goodarzi K, Bendapudi PK, Bornikova L, Gupta S, Leaf DE, Kuter DJ, Rosovsky RP. COVID-19 and coagulation: bleeding and thrombotic manifestations of SARS-CoV-2 infection. Blood. 2020 Jul 23;136(4):489-500. doi: 10.1182/blood.2020006520. PMID 32492712
- [Background] Centers for Disease Control and Prevention. COVID-19 in Racial and Ethnic Minority Groups. 2020.
- [Background] Price-Haywood EG, Burton J, Fort D, Seoane L. Hospitalization and Mortality among Black Patients and White Patients with Covid-19. N Engl J Med. 2020 Jun 25;382(26):2534-2543. doi: 10.1056/NEJMsa2011686. Epub 2020 May 27. PMID 32459916
- [Background] Aldridge RW, Lewer D, Katikireddi SV, Mathur R, Pathak N, Burns R, Fragaszy EB, Johnson AM, Devakumar D, Abubakar I, Hayward A. Black, Asian and Minority Ethnic groups in England are at increased risk of death from COVID-19: indirect standardisation of NHS mortality data. Wellcome Open Res. 2020 Jun 24;5:88. doi: 10.12688/wellcomeopenres.15922.2. eCollection 2020. PMID 32613083
- [Background] Niedzwiedz CL, O'Donnell CA, Jani BD, Demou E, Ho FK, Celis-Morales C, Nicholl BI, Mair FS, Welsh P, Sattar N, Pell JP, Katikireddi SV. Ethnic and socioeconomic differences in SARS-CoV-2 infection: prospective cohort study using UK Biobank. BMC Med. 2020 May 29;18(1):160. doi: 10.1186/s12916-020-01640-8. PMID 32466757
- [Background] Millett GA, Jones AT, Benkeser D, Baral S, Mercer L, Beyrer C, Honermann B, Lankiewicz E, Mena L, Crowley JS, Sherwood J, Sullivan PS. Assessing differential impacts of COVID-19 on black communities. Ann Epidemiol. 2020 Jul;47:37-44. doi: 10.1016/j.annepidem.2020.05.003. Epub 2020 May 14. PMID 32419766
- [Background] Kamin Mukaz D, Gergi M, Koh I, Zakai NA, Judd SE, Sholzberg M, Baumann Kreuziger L, Freeman K, Colovos C, Olson NC, Cushman M. Thrombo-inflammatory biomarkers and D-dimer in a biracial cohort study. Res Pract Thromb Haemost. 2021 Dec 7;5(8):e12632. doi: 10.1002/rth2.12632. eCollection 2021 Dec. PMID 34934895
- [Background] Kosiborod MN, Esterline R, Furtado RHM, Oscarsson J, Gasparyan SB, Koch GG, Martinez F, Mukhtar O, Verma S, Chopra V, Buenconsejo J, Langkilde AM, Ambery P, Tang F, Gosch K, Windsor SL, Akin EE, Soares RVP, Moia DDF, Aboudara M, Hoffmann Filho CR, Feitosa ADM, Fonseca A, Garla V, Gordon RA, Javaheri A, Jaeger CP, Leaes PE, Nassif M, Pursley M, Silveira FS, Barroso WKS, Lazcano Soto JR, Nigro Maia L, Berwanger O. Dapagliflozin in patients with cardiometabolic risk factors hospitalised with COVID-19 (DARE-19): a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet Diabetes Endocrinol. 2021 Sep;9(9):586-594. doi: 10.1016/S2213-8587(21)00180-7. Epub 2021 Jul 21. PMID 34302745
- [Background] Leucker TM, Osburn WO, Reventun P, Smith K, Claggett B, Kirwan BA, de Brouwer S, Williams MS, Gerstenblith G, Hager DN, Streiff MB, Solomon SD, Lowenstein CJ. Effect of Crizanlizumab, a P-Selectin Inhibitor, in COVID-19: A Placebo-Controlled, Randomized Trial. JACC Basic Transl Sci. 2021 Dec;6(12):935-945. doi: 10.1016/j.jacbts.2021.09.013. Epub 2021 Dec 8. PMID 34904132
- [Background] ATTACC Investigators; ACTIV-4a Investigators; REMAP-CAP Investigators; Lawler PR, Goligher EC, Berger JS, Neal MD, McVerry BJ, Nicolau JC, Gong MN, Carrier M, Rosenson RS, Reynolds HR, Turgeon AF, Escobedo J, Huang DT, Bradbury CA, Houston BL, Kornblith LZ, Kumar A, Kahn SR, Cushman M, McQuilten Z, Slutsky AS, Kim KS, Gordon AC, Kirwan BA, Brooks MM, Higgins AM, Lewis RJ, Lorenzi E, Berry SM, Berry LR, Aday AW, Al-Beidh F, Annane D, Arabi YM, Aryal D, Baumann Kreuziger L, Beane A, Bhimani Z, Bihari S, Billett HH, Bond L, Bonten M, Brunkhorst F, Buxton M, Buzgau A, Castellucci LA, Chekuri S, Chen JT, Cheng AC, Chkhikvadze T, Coiffard B, Costantini TW, de Brouwer S, Derde LPG, Detry MA, Duggal A, Dzavik V, Effron MB, Estcourt LJ, Everett BM, Fergusson DA, Fitzgerald M, Fowler RA, Galanaud JP, Galen BT, Gandotra S, Garcia-Madrona S, Girard TD, Godoy LC, Goodman AL, Goossens H, Green C, Greenstein YY, Gross PL, Hamburg NM, Haniffa R, Hanna G, Hanna N, Hegde SM, Hendrickson CM, Hite RD, Hindenburg AA, Hope AA, Horowitz JM, Horvat CM, Hudock K, Hunt BJ, Husain M, Hyzy RC, Iyer VN, Jacobson JR, Jayakumar D, Keller NM, Khan A, Kim Y, Kindzelski AL, King AJ, Knudson MM, Kornblith AE, Krishnan V, Kutcher ME, Laffan MA, Lamontagne F, Le Gal G, Leeper CM, Leifer ES, Lim G, Lima FG, Linstrum K, Litton E, Lopez-Sendon J, Lopez-Sendon Moreno JL, Lother SA, Malhotra S, Marcos M, Saud Marinez A, Marshall JC, Marten N, Matthay MA, McAuley DF, McDonald EG, McGlothlin A, McGuinness SP, Middeldorp S, Montgomery SK, Moore SC, Morillo Guerrero R, Mouncey PR, Murthy S, Nair GB, Nair R, Nichol AD, Nunez-Garcia B, Pandey A, Park PK, Parke RL, Parker JC, Parnia S, Paul JD, Perez Gonzalez YS, Pompilio M, Prekker ME, Quigley JG, Rost NS, Rowan K, Santos FO, Santos M, Olombrada Santos M, Satterwhite L, Saunders CT, Schutgens REG, Seymour CW, Siegal DM, Silva DG Jr, Shankar-Hari M, Sheehan JP, Singhal AB, Solvason D, Stanworth SJ, Tritschler T, Turner AM, van Bentum-Puijk W, van de Veerdonk FL, van Diepen S, Vazquez-Grande G, Wahid L, Wareham V, Wells BJ, Widmer RJ, Wilson JG, Yuriditsky E, Zampieri FG, Angus DC, McArthur CJ, Webb SA, Farkouh ME, Hochman JS, Zarychanski R. Therapeutic Anticoagulation with Heparin in Noncritically Ill Patients with Covid-19. N Engl J Med. 2021 Aug 26;385(9):790-802. doi: 10.1056/NEJMoa2105911. Epub 2021 Aug 4. PMID 34351721
- [Background] REMAP-CAP Investigators; ACTIV-4a Investigators; ATTACC Investigators; Goligher EC, Bradbury CA, McVerry BJ, Lawler PR, Berger JS, Gong MN, Carrier M, Reynolds HR, Kumar A, Turgeon AF, Kornblith LZ, Kahn SR, Marshall JC, Kim KS, Houston BL, Derde LPG, Cushman M, Tritschler T, Angus DC, Godoy LC, McQuilten Z, Kirwan BA, Farkouh ME, Brooks MM, Lewis RJ, Berry LR, Lorenzi E, Gordon AC, Ahuja T, Al-Beidh F, Annane D, Arabi YM, Aryal D, Baumann Kreuziger L, Beane A, Bhimani Z, Bihari S, Billett HH, Bond L, Bonten M, Brunkhorst F, Buxton M, Buzgau A, Castellucci LA, Chekuri S, Chen JT, Cheng AC, Chkhikvadze T, Coiffard B, Contreras A, Costantini TW, de Brouwer S, Detry MA, Duggal A, Dzavik V, Effron MB, Eng HF, Escobedo J, Estcourt LJ, Everett BM, Fergusson DA, Fitzgerald M, Fowler RA, Froess JD, Fu Z, Galanaud JP, Galen BT, Gandotra S, Girard TD, Goodman AL, Goossens H, Green C, Greenstein YY, Gross PL, Haniffa R, Hegde SM, Hendrickson CM, Higgins AM, Hindenburg AA, Hope AA, Horowitz JM, Horvat CM, Huang DT, Hudock K, Hunt BJ, Husain M, Hyzy RC, Jacobson JR, Jayakumar D, Keller NM, Khan A, Kim Y, Kindzelski A, King AJ, Knudson MM, Kornblith AE, Kutcher ME, Laffan MA, Lamontagne F, Le Gal G, Leeper CM, Leifer ES, Lim G, Gallego Lima F, Linstrum K, Litton E, Lopez-Sendon J, Lother SA, Marten N, Saud Marinez A, Martinez M, Mateos Garcia E, Mavromichalis S, McAuley DF, McDonald EG, McGlothlin A, McGuinness SP, Middeldorp S, Montgomery SK, Mouncey PR, Murthy S, Nair GB, Nair R, Nichol AD, Nicolau JC, Nunez-Garcia B, Park JJ, Park PK, Parke RL, Parker JC, Parnia S, Paul JD, Pompilio M, Quigley JG, Rosenson RS, Rost NS, Rowan K, Santos FO, Santos M, Santos MO, Satterwhite L, Saunders CT, Schreiber J, Schutgens REG, Seymour CW, Siegal DM, Silva DG Jr, Singhal AB, Slutsky AS, Solvason D, Stanworth SJ, Turner AM, van Bentum-Puijk W, van de Veerdonk FL, van Diepen S, Vazquez-Grande G, Wahid L, Wareham V, Widmer RJ, Wilson JG, Yuriditsky E, Zhong Y, Berry SM, McArthur CJ, Neal MD, Hochman JS, Webb SA, Zarychanski R. Therapeutic Anticoagulation with Heparin in Critically Ill Patients with Covid-19. N Engl J Med. 2021 Aug 26;385(9):777-789. doi: 10.1056/NEJMoa2103417. Epub 2021 Aug 4. PMID 34351722
- [Background] Berger JS, Kornblith LZ, Gong MN, Reynolds HR, Cushman M, Cheng Y, McVerry BJ, Kim KS, Lopes RD, Atassi B, Berry S, Bochicchio G, de Oliveira Antunes M, Farkouh ME, Greenstein Y, Hade EM, Hudock K, Hyzy R, Khatri P, Kindzelski A, Kirwan BA, Baumann Kreuziger L, Lawler PR, Leifer E, Lopez-Sendon Moreno J, Lopez-Sendon J, Luther JF, Nigro Maia L, Quigley J, Sherwin R, Wahid L, Wilson J, Hochman JS, Neal MD; ACTIV-4a Investigators. Effect of P2Y12 Inhibitors on Survival Free of Organ Support Among Non-Critically Ill Hospitalized Patients With COVID-19: A Randomized Clinical Trial. JAMA. 2022 Jan 18;327(3):227-236. doi: 10.1001/jama.2021.23605. PMID 35040887
- [Derived] Kosiborod MN, Windsor SL, Vardeny O, Berger JS, Reynolds HR, Boumakis S, Althouse AD, Solomon SD, Bhatt AS, Peikert A, Luther JF, Leifer ES, Kindzelski AL, Cushman M, Ng Gong M, Kornblith LZ, Khatri P, Kim KS, Baumann Kreuziger L, Javaheri A, Carpio C, Wahid L, Lopez-Sendon Moreno J, Alonso A, Ho MQ, Lopez-Sendon J, Lopes RD, Curtis JL, Kirwan BA, Geraci MW, Neal MD, Hochman JS; ACTIV-4a Investigators. Effect of sodium-glucose co-transporter-2 inhibitors on survival free of organ support in patients hospitalised for COVID-19 (ACTIV-4a): a pragmatic, multicentre, open-label, randomised, controlled, platform trial. Lancet Diabetes Endocrinol. 2024 Oct;12(10):725-734. doi: 10.1016/S2213-8587(24)00218-3. Epub 2024 Sep 6. PMID 39250922
- [Derived] Greenstein YY, Hubel K, Froess J, Wisniewski SR, Venugopal V, Lai YH, Berger JS, Chang SY, Colovos C, Shah F, Kornblith LZ, Lawler PR, Gaddh M, Guerrero RM, Nkemdirim W, Lopes RD, Reynolds HR, Amigo JS, Wahid L, Zahra A, Goligher EC, Zarychanski R, Leifer E, Huang DT, Neal MD, Hochman JS, Cushman M, Gong MN. Symptoms and Impaired Quality of Life After COVID-19 Hospitalization: Effect of Therapeutic Heparin in Non-ICU Patients in the Accelerating COVID-19 Therapeutic Interventions and Vaccines 4 Acute Trial: Effect on 3-Month Symptoms and Quality of Life. Chest. 2024 Apr;165(4):785-799. doi: 10.1016/j.chest.2023.11.019. Epub 2023 Nov 17. PMID 37979717
- [Derived] Fischer AL, Messer S, Riera R, Martimbianco ALC, Stegemann M, Estcourt LJ, Weibel S, Monsef I, Andreas M, Pacheco RL, Skoetz N. Antiplatelet agents for the treatment of adults with COVID-19. Cochrane Database Syst Rev. 2023 Jul 25;7(7):CD015078. doi: 10.1002/14651858.CD015078. PMID 37489818
- [Derived] Solomon SD, Lowenstein CJ, Bhatt AS, Peikert A, Vardeny O, Kosiborod MN, Berger JS, Reynolds HR, Mavromichalis S, Barytol A, Althouse AD, Luther JF, Leifer ES, Kindzelski AL, Cushman M, Gong MN, Kornblith LZ, Khatri P, Kim KS, Baumann Kreuziger L, Wahid L, Kirwan BA, Geraci MW, Neal MD, Hochman JS; ACTIV4a Investigators. Effect of the P-Selectin Inhibitor Crizanlizumab on Survival Free of Organ Support in Patients Hospitalized for COVID-19: A Randomized Controlled Trial. Circulation. 2023 Aug;148(5):381-390. doi: 10.1161/CIRCULATIONAHA.123.065190. Epub 2023 Jun 25. PMID 37356038
- [Derived] Berger JS, Neal MD, Kornblith LZ, Gong MN, Reynolds HR, Cushman M, Althouse AD, Lawler PR, McVerry BJ, Kim KS, Baumann Kreuziger L, Solomon SD, Kosiborod MN, Berry SM, Bochicchio GV, Contoli M, Farkouh ME, Froess JD, Gandotra S, Greenstein Y, Hade EM, Hanna N, Hudock K, Hyzy RC, Ibanez Estellez F, Iovine N, Khanna AK, Khatri P, Kirwan BA, Kutcher ME, Leifer E, Lim G, Lopes RD, Lopez-Sendon JL, Luther JF, Nigro Maia L, Quigley JG, Wahid L, Wilson JG, Zarychanski R, Kindzelski A, Geraci MW, Hochman JS; ACTIV-4a Investigators. Effect of P2Y12 Inhibitors on Organ Support-Free Survival in Critically Ill Patients Hospitalized for COVID-19: A Randomized Clinical Trial. JAMA Netw Open. 2023 May 1;6(5):e2314428. doi: 10.1001/jamanetworkopen.2023.14428. PMID 37227729
- [Derived] Goligher EC, Lawler PR, Jensen TP, Talisa V, Berry LR, Lorenzi E, McVerry BJ, Chang CH, Leifer E, Bradbury C, Berger J, Hunt BJ, Castellucci LA, Kornblith LZ, Gordon AC, McArthur C, Webb S, Hochman J, Neal MD, Zarychanski R, Berry S, Angus DC; REMAP-CAP, ATTACC, and ACTIV-4a Investigators. Heterogeneous Treatment Effects of Therapeutic-Dose Heparin in Patients Hospitalized for COVID-19. JAMA. 2023 Apr 4;329(13):1066-1077. doi: 10.1001/jama.2023.3651. PMID 36942550
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343
- [Derived] Flumignan RL, Tinoco JDS, Pascoal PI, Areias LL, Cossi MS, Fernandes MI, Costa IK, Souza L, Matar CF, Tendal B, Trevisani VF, Atallah AN, Nakano LC. Prophylactic anticoagulants for people hospitalised with COVID-19. Cochrane Database Syst Rev. 2020 Oct 2;10(10):CD013739. doi: 10.1002/14651858.CD013739. PMID 33502773

RESULTS

PARTICIPANT FLOW:
Groups:
- Therapeutic Dose Anticoagulation: increased dose of heparin above standard of care.
  1.0 - This arm was stopped in severe patients in December 2020 and results are published in PMID: 34351722 (NEJM, August, 2021) (see reference section for citation). This arm was stopped for moderate patients in January 2021.
  theraputic heparin: increased dose of heparin above standard of care.
- Prophylactic Dose Anticoagulation: Heparin standard of care
  1.0 - this arm was stopped for all patients in January, 2021 and results are published in PMID: 34351721 (NEJM, August, 2021) (see reference section for citation)
  prophylactic heparin: standard of care dose of heparin
- Therapeutic Dose Anticoagulation + P2Y12 Inhibitor: increased dose of heparin above standard of care with an added P2Y12 inhibitor
  This Arm enrolled moderate illness patients only. Enrollment of moderate illness patients in the trial was ended per DSMB on June 19, 2021 and results are published in PMID: PMID: 35040887 (JAMA, January, 2022) (see reference section for citation)
  theraputic heparin: increased dose of heparin above standard of care.
  P2Y12: added P2Y12 inhibitor
- Prophylactic Dose Anticoagulation + P2Y12 Inhibitor: Heparin standard of care with an added P2Y12 inhibitor
  This Arm enrolled severe illness patients only. Enrollment of severe illness patients in the trial was ended per DSMB in June 2022.
  prophylactic heparin: standard of care dose of heparin
  P2Y12: added P2Y12 inhibitor
- Standard of Care + SGLT2 Inhibitor: Standard of care plus SGLT2 inhibitor
  This arm will enroll moderate and severe illness patients
  This arm was ended in March 2023
  SGLT2 inhibitor: sglt2 inhibitor
- Standard of Care (SGLT2): Standard of care control for the SLGT2 group
- Standard of Care + Crizanlizumab: Standard of care plus crizanlizumab infusion
  This arm will enroll moderate and severe illness patients
  This arm was ended for all patients per the DSMB in September 2022.
  Crizanlizumab Injection: crizanlizumab injection
- Standard of Care (Criza): Standard of care control for the Criza group
Period: Overall Study
Arm/Group | Therapeutic Dose Anticoagulation | Prophylactic Dose Anticoagulation | Therapeutic Dose Anticoagulation + P2Y12 Inhibitor | Prophylactic Dose Anticoagulation + P2Y12 Inhibitor | Standard of Care + SGLT2 Inhibitor | Standard of Care (SGLT2) | Standard of Care + Crizanlizumab | Standard of Care (Criza)
Started | 569 | 514 | 772 | 739 | 287 | 288 | 211 | 211
Completed | 565 | 511 | 766 | 735 | 280 | 287 | 210 | 209
Not Completed | 4 | 3 | 6 | 4 | 7 | 1 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Standard of Care (SGLT2): This arm will enroll moderate and severe illness patients
  This arm was ended in March 2023
- Standard of Care (Criza): This arm will enroll moderate and severe illness patients
  This arm was ended for all patients per the DSMB in September 2022.
- Total: Total of all reporting groups
Arm/Group | Therapeutic Dose Anticoagulation | Prophylactic Dose Anticoagulation | Therapeutic Dose Anticoagulation + P2Y12 Inhibitor | Prophylactic Dose Anticoagulation + P2Y12 Inhibitor | Standard of Care + SGLT2 Inhibitor | Standard of Care (SGLT2) | Standard of Care + Crizanlizumab | Standard of Care (Criza) | Total
Number analyzed (Participants) | 569 | 514 | 772 | 739 | 287 | 288 | 211 | 211 | 3591
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2
  Between 18 and 65 years | 336 | 300 | 575 | 559 | 57 | 75 | 82 | 61 | 2045
  >=65 years | 233 | 214 | 197 | 178 | 230 | 213 | 129 | 150 | 1544
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 232 | 222 | 295 | 283 | 119 | 123 | 80 | 90 | 1444
  Male | 337 | 292 | 477 | 456 | 168 | 165 | 131 | 121 | 2147
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 12 | 7 | 13 | 17 | 2 | 2 | 1 | 0 | 54
  Asian | 25 | 23 | 20 | 28 | 7 | 14 | 15 | 12 | 144
  Native Hawaiian or Other Pacific Islander | 1 | 2 | 8 | 8 | 1 | 0 | 0 | 1 | 21
  Black or African American | 136 | 89 | 169 | 159 | 37 | 32 | 50 | 48 | 720
  White | 292 | 282 | 455 | 425 | 210 | 201 | 111 | 120 | 2096
  More than one race | 1 | 1 | 5 | 6 | 1 | 0 | 1 | 1 | 16
  Unknown or Not Reported | 102 | 110 | 102 | 96 | 29 | 39 | 33 | 29 | 540
Region of Enrollment [Number; unit: participants]
  United States | 504 | 450 | 574 | 541 | 217 | 219 | 211 | 211 | 2927
  Brazil | 0 | 0 | 88 | 90 | 2 | 3 | 0 | 0 | 183
  Italy | 0 | 0 | 19 | 18 | 2 | 2 | 0 | 0 | 41
  Spain | 65 | 64 | 89 | 86 | 63 | 63 | 00 | 0 | 430
  Mexico | 0 | 0 | 2 | 4 | 3 | 1 | 0 | 0 | 10

OUTCOME MEASURES:

1. Primary Outcome: 21 Day Organ Support (Respiratory or Vasopressor) Free Days
Description: which is defined as the number of days that a patient is alive and free of organ support through the first 21 days after trial entry. Organ Support is defined as receipt of non-invasive mechanical ventilation, high flow nasal canula oxygen, mechanical ventilation, or vasopressor therapy, with death at any time during the index hospitalization assigned -1 days.
  This outcome variable was designed to exceed day 21 on the IQR. It goes above 21 days because it include baseline day 0 in their design.
Time Frame: 21 days from study enrollment
Measure: Median (Inter-Quartile Range); unit: days
Groups:
- Standard of Care (SGLT2): Standard of care for the SGLT2 randomizations
- Standard of Care (Criza): Standard of care for the criza randomizations
Arm/Group | Therapeutic Dose Anticoagulation | Prophylactic Dose Anticoagulation | Therapeutic Dose Anticoagulation + P2Y12 Inhibitor | Prophylactic Dose Anticoagulation + P2Y12 Inhibitor | Standard of Care + SGLT2 Inhibitor | Standard of Care (SGLT2) | Standard of Care + Crizanlizumab | Standard of Care (Criza)
Number analyzed (Participants) | 447 | 462 | 768 | 737 | 285 | 288 | 211 | 210
days | 22 [18 to 22] | 22 [17 to 22] | 17 [1 to 21] | 17 [0 to 21] | 22 [22 to 22] | 22 [22 to 22] | 22 [22 to 22] | 22 [22 to 22]
Statistical Analysis 1: Comparison: Therapeutic Dose Anticoagulation vs Prophylactic Dose Anticoagulation; Test type: Superiority; p = .6778, t-test, 2 sided
Statistical Analysis 2: Comparison: Therapeutic Dose Anticoagulation + P2Y12 Inhibitor vs Prophylactic Dose Anticoagulation + P2Y12 Inhibitor; Test type: Superiority; p = .6292, t-test, 2 sided
Statistical Analysis 3: Comparison: Standard of Care + SGLT2 Inhibitor vs Standard of Care (SGLT2); Test type: Superiority; p = .6858, t-test, 2 sided
Statistical Analysis 4: Comparison: Standard of Care + Crizanlizumab vs Standard of Care (Criza); Test type: Superiority; p = .1351, t-test, 2 sided

2. Secondary Outcome: Death Within 28 Days
Time Frame: 28 days from enrollment
Population: Numbers are different from participant flow due to missing data.
Measure: Count of Participants; unit: Participants
Arm/Group | Therapeutic Dose Anticoagulation | Prophylactic Dose Anticoagulation | Therapeutic Dose Anticoagulation + P2Y12 Inhibitor | Prophylactic Dose Anticoagulation + P2Y12 Inhibitor | Standard of Care + SGLT2 Inhibitor | Standard of Care (SGLT2) | Standard of Care + Crizanlizumab | Standard of Care (Criza)
Number analyzed (Participants) | 450 | 463 | 772 | 739 | 287 | 288 | 211 | 211
Participants | 39 | 52 | 120 | 114 | 37 | 42 | 23 | 13
Statistical Analysis 1: Comparison: Therapeutic Dose Anticoagulation vs Prophylactic Dose Anticoagulation; Test type: Superiority; p = .1959, Chi-squared
Statistical Analysis 2: Comparison: Therapeutic Dose Anticoagulation + P2Y12 Inhibitor vs Prophylactic Dose Anticoagulation + P2Y12 Inhibitor; Test type: Superiority; p = 0.9496, Chi-squared
Statistical Analysis 3: Comparison: Standard of Care + SGLT2 Inhibitor vs Standard of Care (SGLT2); Test type: Superiority; p = .9902, Chi-squared
Statistical Analysis 4: Comparison: Standard of Care + Crizanlizumab vs Standard of Care (Criza); Test type: Superiority; p = .0814, Chi-squared

3. Secondary Outcome: Acute Kidney Injury
Description: Acute Kidney Injury Acute kidney injury after enrollment is defined by KDIGO criteria for Acute Kidney Injury in the setting of not meeting these criteria upon enrollment: Modified Stages: ∙ Stage 2: Serum Cr 2.0-2.9 times baseline ∙ Stage 3: Serum Cr ≥ 3.0 times baseline, OR Increase in serum creatinine to ≥ 4.0mg/dl, OR Initiation of renal replacement therapy
Time Frame: 90 days from enrollment
Population: Analysis was not completed on the Theraputic Dose Anticoagulation or the Prophylactic Dose Anticogulation arms due to not being collected in this protocol. Numbers are different from participant flow due to missing data.
Measure: Count of Participants; unit: Participants
Arm/Group | Therapeutic Dose Anticoagulation | Prophylactic Dose Anticoagulation | Therapeutic Dose Anticoagulation + P2Y12 Inhibitor | Prophylactic Dose Anticoagulation + P2Y12 Inhibitor | Standard of Care + SGLT2 Inhibitor | Standard of Care (SGLT2) | Standard of Care + Crizanlizumab | Standard of Care (Criza)
Number analyzed (Participants) | 0 | 0 | 760 | 733 | 287 | 286 | 188 | 198
Participants | 0 | 0 | 38 | 36 | 5 | 5 | 10 | 10
Statistical Analysis 1: Comparison: Therapeutic Dose Anticoagulation + P2Y12 Inhibitor vs Prophylactic Dose Anticoagulation + P2Y12 Inhibitor; Test type: Superiority; p = 1.0, Chi-squared
Statistical Analysis 2: Comparison: Standard of Care + SGLT2 Inhibitor vs Standard of Care (SGLT2); Test type: Superiority; p = 1, Chi-squared
Statistical Analysis 3: Comparison: Standard of Care + Crizanlizumab vs Standard of Care (Criza); Test type: Superiority; p = 1, Chi-squared

4. Secondary Outcome: Major Thrombotic Event or in Hospital Death
Description: A composite endpoint of death, pulmonary embolism, systemic arterial thromboembolism, myocardial infarction, or ischemic stroke during hospitalization or at 28 days after enrollment (whichever is earlier) - "major thrombotic events or death"
Time Frame: 28 days
Population: Numbers are different from participant flow due to missing data.
Measure: Count of Participants; unit: Participants
Arm/Group | Therapeutic Dose Anticoagulation | Prophylactic Dose Anticoagulation | Therapeutic Dose Anticoagulation + P2Y12 Inhibitor | Prophylactic Dose Anticoagulation + P2Y12 Inhibitor | Standard of Care + SGLT2 Inhibitor | Standard of Care (SGLT2) | Standard of Care + Crizanlizumab | Standard of Care (Criza)
Number analyzed (Participants) | 450 | 463 | 772 | 739 | 287 | 288 | 211 | 211
Participants | 450 | 462 | 174 | 177 | 28 | 33 | 32 | 22
Statistical Analysis 1: Comparison: Therapeutic Dose Anticoagulation vs Prophylactic Dose Anticoagulation; Test type: Superiority; p = .0577, Chi-squared
Statistical Analysis 2: Comparison: Therapeutic Dose Anticoagulation + P2Y12 Inhibitor vs Prophylactic Dose Anticoagulation + P2Y12 Inhibitor; Test type: Superiority; p = .5015, Chi-squared
Statistical Analysis 3: Comparison: Standard of Care + SGLT2 Inhibitor vs Standard of Care (SGLT2); Test type: Superiority; p = .5892, Chi-squared
Statistical Analysis 4: Comparison: Standard of Care + Crizanlizumab vs Standard of Care (Criza); Test type: Superiority; p = .1714, Chi-squared

5. Secondary Outcome: Any Thrombotic Event or in Hospital Death
Description: A composite endpoint of death, pulmonary embolism, systemic arterial thromboembolism, myocardial infarction, DVT, or ischemic stroke during hospitalization or at 28 days after enrollment (whichever is earlier)
Time Frame: 28 days
Population: Numbers are different from participant flow due to missing data.
Measure: Count of Participants; unit: Participants
Arm/Group | Therapeutic Dose Anticoagulation | Prophylactic Dose Anticoagulation | Therapeutic Dose Anticoagulation + P2Y12 Inhibitor | Prophylactic Dose Anticoagulation + P2Y12 Inhibitor | Standard of Care + SGLT2 Inhibitor | Standard of Care (SGLT2) | Standard of Care + Crizanlizumab | Standard of Care (Criza)
Number analyzed (Participants) | 450 | 463 | 772 | 739 | 287 | 288 | 211 | 211
Participants | 450 | 463 | 187 | 177 | 28 | 33 | 32 | 22
Statistical Analysis 1: Comparison: Therapeutic Dose Anticoagulation vs Prophylactic Dose Anticoagulation; Test type: Superiority; p = .0732, Chi-squared
Statistical Analysis 2: Comparison: Therapeutic Dose Anticoagulation + P2Y12 Inhibitor vs Prophylactic Dose Anticoagulation + P2Y12 Inhibitor; Test type: Superiority; p = .9018, Chi-squared
Statistical Analysis 3: Comparison: Standard of Care + SGLT2 Inhibitor vs Standard of Care (SGLT2); Test type: Superiority; p = .5075, Chi-squared
Statistical Analysis 4: Comparison: Standard of Care + Crizanlizumab vs Standard of Care (Criza); Test type: Superiority; p = .1450, Chi-squared

6. Secondary Outcome: Any Renal Replacement Therapy
Time Frame: 28 days
Population: Numbers are different from participant flow due to missing data.
Measure: Count of Participants; unit: Participants
Arm/Group | Therapeutic Dose Anticoagulation | Prophylactic Dose Anticoagulation | Therapeutic Dose Anticoagulation + P2Y12 Inhibitor | Prophylactic Dose Anticoagulation + P2Y12 Inhibitor | Standard of Care + SGLT2 Inhibitor | Standard of Care (SGLT2) | Standard of Care + Crizanlizumab | Standard of Care (Criza)
Number analyzed (Participants) | 450 | 463 | 760 | 733 | 287 | 286 | 188 | 198
Participants | 12 | 12 | 37 | 36 | 1 | 1 | 6 | 4
Statistical Analysis 1: Comparison: Therapeutic Dose Anticoagulation vs Prophylactic Dose Anticoagulation; Test type: Superiority; p = .8837, Chi-squared
Statistical Analysis 2: Comparison: Therapeutic Dose Anticoagulation + P2Y12 Inhibitor vs Prophylactic Dose Anticoagulation + P2Y12 Inhibitor; Test type: Superiority; p = 1, Chi-squared
Statistical Analysis 3: Comparison: Standard of Care + SGLT2 Inhibitor vs Standard of Care (SGLT2); Test type: Superiority; p = 1, Chi-squared
Statistical Analysis 4: Comparison: Standard of Care + Crizanlizumab vs Standard of Care (Criza); Test type: Superiority; p = .5343, Chi-squared

7. Secondary Outcome: Days Free of Organ Support and Renal Replacement Therapy
Description: This outcome variable was designed to exceed day 28 on the IQR. It goes above 28 days because it include baseline day 0 in their design.
Time Frame: 28 days
Population: Numbers are different from participant flow due to missing data.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Therapeutic Dose Anticoagulation | Prophylactic Dose Anticoagulation | Therapeutic Dose Anticoagulation + P2Y12 Inhibitor | Prophylactic Dose Anticoagulation + P2Y12 Inhibitor | Standard of Care + SGLT2 Inhibitor | Standard of Care (SGLT2) | Standard of Care + Crizanlizumab | Standard of Care (Criza)
Number analyzed (Participants) | 447 | 462 | 768 | 737 | 285 | 288 | 211 | 210
days | 29 [25 to 29] | 29 [24 to 29] | 24 [8 to 29] | 24 [2 to 29] | 29 [29 to 29] | 29 [29 to 29] | 29 [29 to 29] | 29 [29 to 29]
Statistical Analysis 1: Comparison: Therapeutic Dose Anticoagulation vs Prophylactic Dose Anticoagulation; Test type: Superiority; p = .6636, t-test, 2 sided
Statistical Analysis 2: Comparison: Therapeutic Dose Anticoagulation + P2Y12 Inhibitor vs Prophylactic Dose Anticoagulation + P2Y12 Inhibitor; Test type: Superiority; p = .5878, t-test, 2 sided
Statistical Analysis 3: Comparison: Standard of Care + SGLT2 Inhibitor vs Standard of Care (SGLT2); Test type: Superiority; p = .7148, t-test, 2 sided
Statistical Analysis 4: Comparison: Standard of Care + Crizanlizumab vs Standard of Care (Criza); Test type: Superiority; p = .1117, t-test, 2 sided

8. Secondary Outcome: Ventilator Free Days up to Day 28
Description: as for outcome 7
Time Frame: 28 days
Population: Numbers are different from participant flow due to missing data.
Measure: Mean (Inter-Quartile Range); unit: days
Arm/Group | Therapeutic Dose Anticoagulation | Prophylactic Dose Anticoagulation | Therapeutic Dose Anticoagulation + P2Y12 Inhibitor | Prophylactic Dose Anticoagulation + P2Y12 Inhibitor | Standard of Care + SGLT2 Inhibitor | Standard of Care (SGLT2) | Standard of Care + Crizanlizumab | Standard of Care (Criza)
Number analyzed (Participants) | 447 | 462 | 768 | 737 | 285 | 288 | 211 | 210
days | 24.89 [29 to 29] | 24.63 [29 to 29] | 21.09 [14 to 29] | 20.83 [10 to 29] | 26.22 [29 to 29] | 26.42 [29 to 29] | 25.32 [29 to 29] | 26.69 [29 to 29]
Statistical Analysis 1: Comparison: Therapeutic Dose Anticoagulation vs Prophylactic Dose Anticoagulation; Test type: Superiority; p = .6780, t-test, 2 sided
Statistical Analysis 2: Comparison: Therapeutic Dose Anticoagulation + P2Y12 Inhibitor vs Prophylactic Dose Anticoagulation + P2Y12 Inhibitor; Test type: Superiority; p = .6638, t-test, 2 sided
Statistical Analysis 3: Comparison: Standard of Care + SGLT2 Inhibitor vs Standard of Care (SGLT2); Test type: Superiority; p = .7645, t-test, 2 sided
Statistical Analysis 4: Comparison: Standard of Care + Crizanlizumab vs Standard of Care (Criza); Test type: Superiority; p = 0.0987, t-test, 2 sided

9. Secondary Outcome: Days Free of Vasopressors
Description: as for outcome 7
Time Frame: 28 days
Population: Numbers are different from participant flow due to missing data.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Therapeutic Dose Anticoagulation | Prophylactic Dose Anticoagulation | Therapeutic Dose Anticoagulation + P2Y12 Inhibitor | Prophylactic Dose Anticoagulation + P2Y12 Inhibitor | Standard of Care + SGLT2 Inhibitor | Standard of Care (SGLT2) | Standard of Care + Crizanlizumab | Standard of Care (Criza)
Number analyzed (Participants) | 447 | 462 | 768 | 737 | 285 | 288 | 211 | 210
days | 29 [29 to 29] | 29 [29 to 29] | 29 [26 to 29] | 29 [25 to 29] | 29 [29 to 29] | 29 [29 to 29] | 29 [29 to 29] | 29 [29 to 29]
Statistical Analysis 1: Comparison: Therapeutic Dose Anticoagulation vs Prophylactic Dose Anticoagulation; Test type: Superiority; p = .4016, t-test, 2 sided
Statistical Analysis 2: Comparison: Therapeutic Dose Anticoagulation + P2Y12 Inhibitor vs Prophylactic Dose Anticoagulation + P2Y12 Inhibitor; Test type: Superiority; p = .5815, t-test, 2 sided
Statistical Analysis 3: Comparison: Standard of Care + SGLT2 Inhibitor vs Standard of Care (SGLT2); Test type: Superiority; p = .9085, t-test, 2 sided
Statistical Analysis 4: Comparison: Standard of Care + Crizanlizumab vs Standard of Care (Criza); Test type: Superiority; p = .0820, t-test, 2 sided

10. Secondary Outcome: Progression to Intubation or Death
Description: analysis completed on the Heparin protocol
Time Frame: 28 days
Population: Numbers are different from participant flow due to missing data.
Measure: Count of Participants; unit: Participants
Arm/Group | Therapeutic Dose Anticoagulation | Prophylactic Dose Anticoagulation | Therapeutic Dose Anticoagulation + P2Y12 Inhibitor | Prophylactic Dose Anticoagulation + P2Y12 Inhibitor | Standard of Care + SGLT2 Inhibitor | Standard of Care (SGLT2) | Standard of Care + Crizanlizumab | Standard of Care (Criza)
Number analyzed (Participants) | 450 | 463 | 770 | 737 | 280 | 283 | 210 | 205
Participants | 450 | 463 | 768 | 735 | 273 | 278 | 209 | 199
Statistical Analysis 1: Comparison: Therapeutic Dose Anticoagulation vs Prophylactic Dose Anticoagulation; Test type: Superiority; p = .3135, Chi-squared
Statistical Analysis 2: Comparison: Therapeutic Dose Anticoagulation + P2Y12 Inhibitor vs Prophylactic Dose Anticoagulation + P2Y12 Inhibitor; Test type: Superiority; p = .9581, Chi-squared
Statistical Analysis 3: Comparison: Standard of Care + SGLT2 Inhibitor vs Standard of Care (SGLT2); Test type: Superiority; p = .9661, Chi-squared
Statistical Analysis 4: Comparison: Standard of Care + Crizanlizumab vs Standard of Care (Criza); Test type: Superiority; p = .1073, Chi-squared

11. Secondary Outcome: Survival Until Discharge
Time Frame: 28 days
Population: Numbers are different from participant flow due to missing data.
Measure: Count of Participants; unit: Participants
Arm/Group | Therapeutic Dose Anticoagulation | Prophylactic Dose Anticoagulation | Therapeutic Dose Anticoagulation + P2Y12 Inhibitor | Prophylactic Dose Anticoagulation + P2Y12 Inhibitor | Standard of Care + SGLT2 Inhibitor | Standard of Care (SGLT2) | Standard of Care + Crizanlizumab | Standard of Care (Criza)
Number analyzed (Participants) | 450 | 463 | 772 | 739 | 287 | 288 | 211 | 211
Participants | 406 | 409 | 633 | 598 | 264 | 266 | 186 | 197
Statistical Analysis 1: Comparison: Therapeutic Dose Anticoagulation vs Prophylactic Dose Anticoagulation; Test type: Superiority; p = .3575, Chi-squared
Statistical Analysis 2: Comparison: Therapeutic Dose Anticoagulation + P2Y12 Inhibitor vs Prophylactic Dose Anticoagulation + P2Y12 Inhibitor; Test type: Superiority; p = .5910, Chi-squared
Statistical Analysis 3: Comparison: Standard of Care + SGLT2 Inhibitor vs Standard of Care (SGLT2); Test type: Superiority; p = .8670, Chi-squared
Statistical Analysis 4: Comparison: Standard of Care + Crizanlizumab vs Standard of Care (Criza); Test type: Superiority; p = .0645, Chi-squared

ADVERSE EVENTS:
Time Frame: Discharge, Death or Day 28
Description: Non Serious adverse events were not collected.
Groups:
- Standard of Care (sglt2): Standard of care for sglt2 randomzations
  This arm will enroll moderate and severe illness patients
- Standard of Care (Criza): Standard of care for criza randomizations
  This arm will enroll moderate and severe illness patients
Arm/Group | Therapeutic Dose Anticoagulation | Prophylactic Dose Anticoagulation | Therapeutic Dose Anticoagulation + P2Y12 Inhibitor | Prophylactic Dose Anticoagulation + P2Y12 Inhibitor | Standard of Care + SGLT2 Inhibitor | Standard of Care (sglt2) | Standard of Care + Crizanlizumab | Standard of Care (Criza)
All-Cause Mortality (participants affected / at risk) | 69/569 | 65/514 | 147/772 | 149/739 | 37/287 | 42/288 | 37/211 | 28/211
Serious Adverse Events (participants affected / at risk) | 46/569 | 57/514 | 151/772 | 133/739 | 20/287 | 33/288 | 24/211 | 28/211
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Therapeutic Dose Anticoagulation (N=569) | Prophylactic Dose Anticoagulation (N=514) | Therapeutic Dose Anticoagulation + P2Y12 Inhibitor (N=772) | Prophylactic Dose Anticoagulation + P2Y12 Inhibitor (N=739) | Standard of Care + SGLT2 Inhibitor (N=287) | Standard of Care (sglt2) (N=288) | Standard of Care + Crizanlizumab (N=211) | Standard of Care (Criza) (N=211)
Deep Vein Thrombosis (Vascular disorders) | 1 | 2 | 1 | 0 | 0 | 3 | 1 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 10 | 18 | 41 | 26 | 2 | 3 | 0 | 4
myocardial infarction (Cardiac disorders) | 2 | 2 | 7 | 4 | 0 | 1 | 2 | 1
ischemmic stroke (Vascular disorders) | 3 | 3 | 11 | 3 | 0 | 1 | 0 | 0
Other arterial or venous thromboembolism event (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
disseminated intravascular coagulation (Vascular disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
symptomatic intracranial or intracerebral hemorrhage (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
major bleeding (Vascular disorders) | 13 | 8 | 21 | 17 | 4 | 3 | 6 | 4
heparin induced thrombocytopenia (Injury, poisoning and procedural complications) | 2 | 3 | 3 | 3 | 0 | 0 | 0 | 0
diabetic ketoacidosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
acute kidney injury (Renal and urinary disorders) | 0 | 0 | 3 | 0 | 4 | 7 | 9 | 10
anaphylaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
other (Injury, poisoning and procedural complications) | 2 | 3 | 24 | 34 | 9 | 8 | 4 | 1
arterial thromboembolic event (Vascular disorders) | 2 | 2 | 0 | 2 | 0 | 1 | 0 | 2
Venus thrombosis (Vascular disorders) | 10 | 14 | 47 | 47 | 1 | 5 | 4 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2021-10-19): https://cdn.clinicaltrials.gov/large-docs/74/NCT04505774/Prot_001.pdf
  • Statistical Analysis Plan (2021-06-04): https://cdn.clinicaltrials.gov/large-docs/74/NCT04505774/SAP_003.pdf
  • Informed Consent Form (2021-10-22): https://cdn.clinicaltrials.gov/large-docs/74/NCT04505774/ICF_000.pdf